CLINICAL TRIAL: NCT02893475
Title: Impact de la durée de Dialyse Avant Greffe rénale Avec Donneur Vivant Sur la qualité de Vie et la réinsertion Professionnelle Des Receveurs
Brief Title: Impact of Preemptive Living Donor Renal Transplantation on Quality of Life , Occupational Rehabilitation and Societal Participation of Transplant Recipients
Acronym: QUAVIREIN_RDDV
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: Quavirein_RDDV1
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Living donor (LD) kidney transplantation is currently the best treatment for end-stage renal disease (ESRD) in terms of life expectancy and quality of life. This method allows preemptive transplantation, before beginning dialysis.

The main objective of this study will be to investigate quality of life and societal participation in a population of LD kidney transplant recipients comparing preemptive LD transplantation versus non-preemptive transplantation (performed after a period of dialysis).

DETAILED DESCRIPTION:
Living donor (LD) kidney transplantation is currently the best treatment for end-stage renal disease (ESRD) in terms of life expectancy and quality of life. This method allows preemptive transplantation, before beginning dialysis.

The main objective of this study will be to investigate quality of life and societal participation in a population of LD kidney transplant recipients comparing preemptive LD transplantation versus non-preemptive transplantation (performed after a period of dialysis).

It is hypothesized that in addition to prolonged graft survival, preemptive LD kidney transplantation is associated with less deterioration of quality of life and better societal participation.

We therefore propose a cross-sectional population-based study to include all patients who underwent LD kidney transplantation from 2004 through 2009 in the seven most active kidney transplantation centers in France. Cross-sectional surveys have been conducted since 2004 by the biomedicine agency in collaboration with the InVS in order to evaluate quality of life among ESRD patients. The most recent survey, QUAVIREIN, is in process but has included only a small number of patients selected at random. We want to broaden the study population beyond the QUAVIREIN sample in order to include the entire population of LD kidney transplant recipients.

The study population will thus include all patients who received a LD kidney transplant from 2004 through 2009 who give their informed consent to participate in the study and have a functional transplant on March 31, 2012. The seven transplantation centers have agreed to participate in the study.

The patients will be identified using the CRISTAL and QUAVIREIN databases. Quality of life, occupational rehabilitation and societal participation data will be collected with a self-administered questionnaire sent to all identified patients, excepting (in order to avoid duplicates) those who have already participated in the QUAVIREIN survey. The methodology and data collection will be the same as for QUAVIREIN. The Department of Epidemiology and Clinical Evaluation (CIC-EC) of the Nancy University Hospital Center will be in charge of the study logistics and organization.

The study hypothesis will be tested by applying univariate then multivariate statistical analysis to the collected data using ad hoc models comparing preemptive transplantation versus non-preemptive transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* LD kidney transplantation from 2004 through 2009
* First LD kidney transplantation in the seven most active kidney transplantation centers in France: Paris Necker, Nancy, Paris Saint Louis, Foch, Nantes, Toulouse and Montpellier
* Patient with a functioning kidney at the time of the study
* Patient able to read and understand French

Exclusion Criteria:

* Patient with multiple transplantation including liver transplantation
* Patient unable to read and understand French
* Patient died or lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population-based
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Quality of life | through study completion, an average of 1 year
  SF-36 and Retransqol questionnaires

SECONDARY OUTCOMES:
Societal participation | through study completion, an average of 1 year
  self-administered questionnaire
Professional reintegration | through study completion, an average of 1 year
  self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ayav, MD, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No